CLINICAL TRIAL: NCT04458103
Title: Percutaneous RVAD to Preemptively Treat Right Heart Failure Post-LVAD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: There were excess adverse events in study population compared to baseline controls
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David A. D'Alessandro, M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020P000422
Record Dates: First submitted 2020-06-16; First posted 2020-07-07 (Actual); Results first posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- prospective interventional cohort (Experimental): The prospective interventional cohort will consist of patients undergoing LVAD implantation at Massachusetts General Hospital. These patients will receive an RVAD (either the ProtekDuo or Impella RP) prior to or during LVAD implantation.
  Interventions: Device: Percutaneous RVAD
- retrospective control cohort (No Intervention): The historical control cohort will consist of retrospective data collection on patients who have undergone LVAD implantation in the past. This group will be age and sex matched with the enrolled prospective interventional patients.

INTERVENTIONS:
Device: Percutaneous RVAD — ProtekDuo or Impella RP
  Arms: prospective interventional cohort

SUMMARY:
Prior studies have shown that left ventricular assist device (LVAD) implantation commonly results in right ventricular failure (RVF). Right ventricular dysfunction and failure after LVAD implantation is known to increase morbidity and mortality and contribute to longer post-implant hospital length of stay. Since RVF is difficult to predict and can have harmful effects such as increased ICU stay, adverse outcomes, and mortality, it could be beneficial to preemptively treat patients through preoperative or intraoperative percutaneous right ventricular assist device (RVAD) placement to prevent RVF.

This trial will include both a prospective interventional cohort and a retrospective control cohort. The prospective interventional cohort will consist of patients undergoing LVAD implantation at Massachusetts General Hospital. These patients will preemptively receive an RVAD (either the ProtekDuo or Impella RP) surrounding LVAD implantation. The historical control cohort will consist of retrospective data collection on patients who have undergone LVAD implantation in the past. This group will be matched with the enrolled prospective interventional patients. The purpose of this study is to compare clinical outcomes of standard of care treatment versus percutaneous RVAD placement perioperatively to LVAD implantation. The investigators hypothesize that the use of the RVAD will mitigate need for inotropic support, reducing the vasoactive-inotrope score (VIS) by 50%, and will improve end organ function in patients compared to standard of care.

Subjects who consent to the study will undergo peri-operative placement of an RVAD, which will be left in up to 72 hours postoperatively. The type of RVAD (Impella RP or ProtekDuo) inserted will be determined by patient needs and venous access and will be up to the discretion of the treating physician. 25 subjects will be enrolled in the prospective interventional cohort and compared to 25 subjects in the matched retrospective control cohort.

DETAILED DESCRIPTION:
Prior studies have shown that left ventricular assist device (LVAD) implantation commonly results in right ventricular failure (RVF). Right ventricular dysfunction and failure after LVAD implantation is known to increase morbidity and mortality and contribute to longer post-implant hospital length of stay. More severe right ventricular failure is highly correlated with poor prognosis and death post-LVAD implantation. In current practice, patients who receive LVADs require right heart support, provided in the form of inotropes. Vasoactive inotrope score (VIS) is a measure that quantifies the amount of right heart support required post-operatively, including dopamine, dobutamine, milrinone, epinephrine, norepinephrine, and vasopressin. It has been used in other studies as a surrogate marker for hemodynamic cardiovascular derangement.

In some cases, right ventricular failure post-LVAD also requires mechanical circulatory support during the perioperative period. Since RVF is difficult to predict and can have harmful effects such as increased ICU stay, adverse outcomes, and mortality, it could be beneficial to preemptively treat patients through preoperative or intraoperative percutaneous right ventricular assist device (RVAD) placement to prevent RVF. The purpose of this study is to test the hypothesis that preemptive use of percutaneous RVADs will mitigate the need for inotropic support in LVAD patients, reducing associated adverse outcomes.

This trial will include both a prospective interventional cohort and a retrospective control cohort. The prospective interventional cohort will consist of patients undergoing LVAD implantation at Massachusetts General Hospital. These patients will receive an RVAD (either the ProtekDuo or Impella RP) prior to or during LVAD implantation. The historical control cohort will consist of retrospective data collection on patients who have undergone LVAD implantation in the past. This group will be matched with the enrolled prospective interventional patients. The purpose of this study is to compare clinical outcomes of standard of care treatment versus preemptive percutaneous RVAD placement surrounding LVAD implantation. The investigators hypothesize that the use of the RVAD will mitigate need for inotropic support, reducing the vasoactive-inotrope score (VIS) by 50%, and will improve end organ function in patients compared to standard of care.

There are two types of percutaneous RVADs that will be used in the study: the Impella RP and the ProtekDuo. These devices allow for early intervention in RVF without the need for invasive surgical procedures requiring placement of durable RVADs via thoracotomy or sternotomy. The Impella RP, manufactured by Abiomed, is a heart pump that delivers blood from the inferior vena cava (IVC) to the pulmonary artery (PA). Its insertion is done percutaneously via catheterization through the femoral vein. ProtekDuo, manufactured by TandemLife, is another device placed percutaneously for right heart support via the right internal jugular (RIJ) vein.

Subjects who consent to the study will undergo pre-operative or intra-operative placement of an RVAD, which will be left in up to 72 hours postoperatively. The type of RVAD (Impella RP or ProtekDuo) inserted will be determined by patient needs and venous access and will be up to the discretion of the treating physician. 25 subjects will be enrolled in the prospective interventional cohort and compared to 25 subjects in the matched retrospective control cohort.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-75
* Accepted for LVAD implantation by MGH multidisciplinary team

Exclusion Criteria:

* Disorders of the pulmonary artery wall that would preclude placement or correct positioning of RVAD
* Presence of mechanical valves
* Mural thrombosis of the right atrium or vena cava
* Anatomic conditions precluding insertion of the RVAD
* Complicated venous access precluding or complicating device placement (i.e. femoral and jugular thrombosis)
* No evidence of right ventricular dysfunction by echocardiogram

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prospective Interventional Cohort | Retrospective Control Cohort
Started | 17 | 144
Completed | 17 | 144
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prospective Interventional Cohort | Retrospective Control Cohort | Total
Number analyzed (Participants) | 17 | 144 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.41 (13.97) | 58.13 (13.31) | 58.3 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 34 | 38
  Male | 13 | 110 | 123
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 15 | 16
  White | 12 | 111 | 123
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 14 | 16
Region of Enrollment [Number; unit: participants]
  United States | 17 | 144 | 161

OUTCOME MEASURES:

1. Primary Outcome: Vasoactive Inotropic Score
Description: Retrospective review in a patient chart. Score calculated based on dosages of vasopressors and inotropes within first 24-hours post-LVAD implant. The maximum Vasoactive Inotropic Score within the first 24-hours is reported.
  Vasoactive Inotropic Score= dopamine (μg/kg/min) + dobutamine (μg/kg/min) + 10 x milrinone (μg/kg/min) + 100 x epinephrine (μg/kg/min) + 100 x norepinephrine (μg/kg/min) + 10,000 x vasopressin (U/kg/min).
  Minimum possible vasoactive inotropic score is 0. It is hypothesized that a higher score will correspond with worse outcomes.
Time Frame: first 24 hours post-LVAD implantation
Measure: Mean (Standard Deviation); unit: Vasoactive Inotropic Score
Arm/Group | Prospective Interventional Cohort | Retrospective Control Cohort
Number analyzed (Participants) | 17 | 144
Vasoactive Inotropic Score | 36.4 (103.1) | 47.46 (84.8)

2. Secondary Outcome: Intensive Care Unit Length of Stay
Description: Retrospective review in a patient chart
Time Frame: up to date of discharge from intensive care unit (estimated average = 1 week)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Prospective Interventional Cohort | Retrospective Control Cohort
Number analyzed (Participants) | 17 | 144
days | 14.1 (14.9) | 11.1 (13.7)

3. Secondary Outcome: Total Post-operative Length of Stay After LVAD Implantation
Description: Retrospective review in a patient chart
Time Frame: up to date of hospital discharge (estimated average = 3 weeks)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Prospective Interventional Cohort | Retrospective Control Cohort
Number analyzed (Participants) | 17 | 144
days | 30.2 (31.1) | 24.9 (17.8)

4. Secondary Outcome: Survival at Discharge After LVAD Placement
Description: Retrospective review in a patient chart
Time Frame: up to date of hospital discharge (estimated average = 3 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective Interventional Cohort | Retrospective Control Cohort
Number analyzed (Participants) | 17 | 144
Participants | 13 | 139

5. Secondary Outcome: Survival at 1 Year After LVAD Placement or Heart Transplant
Description: Retrospective review in a patient chart
Time Frame: up to 1 year post-LVAD implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective Interventional Cohort | Retrospective Control Cohort
Number analyzed (Participants) | 17 | 144
Participants | 13 | 139

6. Secondary Outcome: End Organ Dysfunction
Description: end organ dysfunction including 1) Development of acute kidney injury (AKI) - defined as increase in serum creatinine (sCr) to 4mg/dl or greater, a 150 percent or greater increase in sCr over the baseline preoperative value, or a new requirement for renal replacement therapy
Time Frame: up to 1 year post-LVAD implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective Interventional Cohort | Retrospective Control Cohort
Number analyzed (Participants) | 17 | 144
Participants | 5 | 27

ADVERSE EVENTS:
Time Frame: 1year
Description: INTERMACS Adverse Event Definitions
Arm/Group | Prospective Interventional Cohort | Retrospective Control Cohort
All-Cause Mortality (participants affected / at risk) | 4/17 | 13/144
Serious Adverse Events (participants affected / at risk) | 16/17 | 135/144
Other Adverse Events (participants affected / at risk) | 8/17 | 74/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prospective Interventional Cohort (N=17) | Retrospective Control Cohort (N=144)
Bleed (Blood and lymphatic system disorders) | 6 | 56
Neurological Event (Nervous system disorders) | 3 | 13
Infection (Infections and infestations) | 7 | 66
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prospective Interventional Cohort (N=17) | Retrospective Control Cohort (N=144)
Renal Dysfunction (Renal and urinary disorders) | 5 | 27
Arrhythmia (Cardiac disorders) | 5 | 46
Respiratory Dysfunction (Respiratory, thoracic and mediastinal disorders) | 5 | 25
Hepatic Dysfunction (Hepatobiliary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/03/NCT04458103/Prot_002.pdf
  • Statistical Analysis Plan (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/03/NCT04458103/SAP_003.pdf